CLINICAL TRIAL: NCT02418377
Title: Whole-exome Sequencing to Identify Genetic Variants Associated With Severe Childhood Obesity, and Tracking the Changing Prevalence of Obesity Related Complications
Brief Title: Whole-exome Sequencing in Childhood Obesity
Status: Completed | Type: Observational
Sponsor: National University of Singapore (Other)
Collaborators: Health Promotion Board, Singapore (Other Government); Genome Institute of Singapore (Other)
Responsible Party: Principal Investigator, Lee Yung Seng, Professor, National University of Singapore
Other Study IDs: NMRC/CIRG/1407/2014
Record Dates: First submitted 2015-04-12; First posted 2015-04-16 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Childhood Obesity
Keywords: Obesity; Genetics; Whole exome sequencing; Children
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples With DNA — 15-19mls of blood will be extracted from each subject. Blood will be processed to obtain plasma/serum and DNA will be extracted from blood cells.
  Plasma/serum and DNA samples will be stored at -80degree Celsius.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese children: The obese subject must meet all of the following inclusion criteria to participate in this study:
  1. Ideal body weight for height (WFH) of at least 140% or BMI for age above 97th percentile
  2. Overweight before 10 years of age
  3. Informed consent from both obese children subject and legal representative e.g. parents
- Family members of obese children: Family member must meet all of the following inclusion criteria to participate in this study:
  1. Must be parent or direct sibling of obese subject
  2. Informed consent from both subject and parent is subject is below 21 years of age

SUMMARY:
Obesity is a complex multifactorial disease where genetics play an important role in predisposing children to early onset obesity. Though many obesity susceptible genes and variants have been identified with obesity, the most common obesity gene, MC4R only accounts for 5% of all early onset obesity cases. This implies that there may be more obesity related genes and variants that need to be unravelled to further delineate the relationship between obesity and genetics. The investigators propose in screening the exonic regions of all the genes in obese subjects using whole-exome sequencing (WES) to discover novel obesity related variants and genes.

Primary hypothesis The investigators hypothesized that our paediatric subjects with early-onset severe obesity will have strong genetic predisposition and therefore the cohort would be enriched with obesity susceptibility genetic variants.

Secondary hypothesis The investigators hypothesized that there is increasing prevalence of, and possibly worsening, obesity-related complications (namely glucose intolerance, hypertension, metabolic syndrome, non-alcoholic fatty liver disease) in our severely obese children, as compared to 15 years ago, due to an increasingly obesogenic environment promoting unhealthy lifestyle and eating habits.

DETAILED DESCRIPTION:
Number of subjects to be enrolled:

As our study aims to identify susceptible genetic variants associated with early onset obesity, we will be recruiting 400 obese children to participate in this genetic study, in addition to the existing DNA samples we collected in a previous study (DSRB Ref C/00/501). These 400 obese children will be recruited through NUH paediatric clinic and School Health Clinic at Health Promotion Board. We will also recruit family members of the obese children who are interested to join the research study. We will be using the DNA samples and information of 250 obese children previously recruited to the Obesity Genetic Study from January 2000 to December 2004 (DSRB Ref C/00/501). We will also be performing WES on 500 lean adults (as controls) recruited for an ongoing study titled "Whole exome sequencing to identify genes for extreme Myopia in Asian populations" (NUS-IRB reference code: 12-466).

Total number of new obese children subjects to be recruited: 400 Total number of family members (Parents and siblings): 500 Total number of existing obese children subjects to be used: 250 Total number of existing lean adult controls to be used: 500

Criteria for Recruitment:

The doctor will ask a few simple questions regarding the age and medical history of subjects.

For obese subjects: Overweight before 10 years of age, and the body weight is 40% above the ideal body weight for height, or BMI for age above 97th percentile without any major medical illness.

For family members: Parents or direct siblings of obese children (no selection criteria) For controls: Lean adults of ongoing study (NUS-IRB reference code: 12-466) with BMI between 18.5 kg/m2 and 23 kg/m2

Inclusion Criteria:

The obese subject must meet all of the following inclusion criteria to participate in this study:

1. Ideal body weight for height (WFH) of at least 140% or BMI for age above 97th percentile
2. Overweight before 10 years of age
3. Informed consent from both obese children subject and legal representative e.g. parents

Family member must meet all of the following inclusion criteria to participate in this study:

1. Must be parent or direct sibling of obese subject
2. Informed consent from both subject and parent is subject is below 21 years of age

Exclusion Criteria:

All subjects meeting any of the exclusion criteria at baseline will be excluded from participation:

1. Unfit for blood testing and OGTT testing
2. No informed consent

Withdrawal Criteria:

The study may be discontinued if:

* No OSHE approval
* No DSRB approval
* Complaints of any inappropriate procedures performed on subjects
* Laboratory toxicity

Study Visits and Procedures:

1. Screening Visits and Procedures The subject will be screened at the school health clinic at HPB or NUH paediatric clinic. The subject's age, weight and height will be taken. Only those who the doctor determined to have an ideal body weight for height of greater than 140% or BMI for age at greater than 97th percentile of the local children population will be invited for the study. The subject will be allowed to go home with the consent form and reply within 3 months before recruitment.
2. Study Visits and Procedures Study visit 1: Trained doctor will carry out an interview regarding the medical history if the subject and performed physical examination. 15ml of blood will be drawn from the subject (after overnight fasting) for testing of liver panel, lipid panel, fasting insulin level, fasting C-peptide level. The subject will also go through an oral glucose tolerance test (OGTT) where 2ml of blood will be drawn at both 0 min and 120min time-interval during OGTT. During the 2 hr OGTT, the subjects will be required to fill in 3 sets of questionnaire regarding motivational level, socio-economic status and physical activity and diet.

   The family member of the obese subject is required to go through all testing as described above for the subject except that they do not need to undergo OGTT.
3. Final Study Visit:

   The final study visit will be scheduled 2-3 weeks after the first visit. The screening report of the subject will be reviewed and evaluated by the attending doctor to the subject.
4. Post Study Follow up and Procedures The subject will be able to keep a copy of their health screening test reports. For subjects who are found to suffer from medical conditions such as dyslipidemia, high blood pressure, high body fat percentage, liver malfunction or glucose intolerance, they will be referred to other departments for further testing and medical attention to confirm outcome measures. Subjects found to have a rare genetic variant through genetic testing will also be called back for further and repeat clinical examination and testing.
5. Discontinuation Visit and Procedures Subjects may withdraw voluntarily from participation in the study at any time. The biological samples of the subject will be discarded upon the request of the subject. However, if the patient was found to be suffering from any other complications during the study health screening, they will be advised and referred to other departments for medical treatment.

Data Quality Assurance:

The electronic input of patients' data into the system will be handled by 2 research coordinators who will perform the data entry independently. Thus, data of each subject will be entered twice into the system by the 2 independent research coordinators. We will do a system comparison between the 2 entries for per subject to ensure that all information of the subject was entered correctly and accurately. The principal investigator will also randomly check through the system every month for data quality assurance.

Data Entry and Storage:

The clinical testing data and questionnaire will be entered by the subjects on paper. The paper documentations will be transferred or transported back to the PI's office and each subject's data will be entered electronically by 2 independent research coordinators to ensure data quality assurance. All electronic entry of the documentations can only be performed within the office using the office computer and all paper documentations must be returned for lock-up at the end of the day. The electronic documentations will be password protected and the hard copy of the paper documentations will be stored in a lock and key access cabinet in PI's office. Briefly discuss where data will be entered (i.e. will these entries be on paper or electronically), stored and handled.

Determination of Sample Size:

Power calculations were carried out using Quanto (ver 1.2.4). To detect variants at a power of odd ratios of 2.0-5.0 in the discovery stage at varying MAF (α=0.01), the sample size of 400 obese children is approximately 51% to 98% power to detect variants with large effects (OR = 3.5) in our discovery stage, at MAF between 0.5% and 3.0%, respectively (α=0.01).

Statistical and Analytical Plans:

All prioritized damaging non-synonymous variants will be tested for statistical association in a case-control design using SPSS. The 2-tailed Fisher's exact test will be utilized for variants with MAF < 3% and logistic regression, adjusting for sex will be performed for variants with MAF ≥ 3%. These will be done using PLINK. We will also carry out a gene-level burden tests using the Sequencing Kernel Association Test (SKAT) software. All single-variant and gene-level results will be corrected for multiple tests using a Bonferonni correction. Any variants identified by prediction tool (Polyphen2) to be highly disruptive (defined as nonsense, splice site and frameshift changes, which severely disrupt protein structure) will be prioritized for validations.

Statistical analyses of de novo genotyping data will be similar to that in primary aim 1. Subsequently, we will meta-analyse data from the discovery and validation stages using an inverse variance-weighted method, assuming a fixed-effect model, to derive overall pooled estimates and two-sided p-values. Heterogeneity checks will be conducted (Cochran's Q and I2 indices), and at variants where significant (Q p-value <0.05 and/or I2 index >40%) heterogeneity is detected the meta-analysis will be carried out in the random effects mode as well.

RETENTION OF TRIAL DOCUMENTS:

The records for all participants which include the medical history, clinical report, blood test results, questionnaire, OSHE documentation, IRB documentation and DSRB documentation will be kept by the principal investigator in a lock-up cabinet in his card access office. Only the principal investigator will hold the key and have direct access to the lock-up cabinet. These documents will be retained for a period of 6years after the end of the research study.

For Principal Investigator initiated Trials:

All serious adverse events (SAEs) that are unexpected and related to the study drug must be reported to HSA.

"A serious adverse event or serious adverse drug reaction is any untoward medical occurrence at any dose that:

* Results in death.
* Is life-threatening (immediate risk of death).
* Requires inpatient hospitalization or prolongation of existing hospitalization.
* Results in persistent or significant disability/incapacity.
* Results in congenital anomaly/birth defect.
* Is a Medically important event.

Medical and scientific judgment should be exercised in determining whether an event is an important medical event. An important medical event may not be immediately life threatening and/or result in death or hospitalization. However, if it is determined that the event may jeopardize the subject and/or may require intervention to prevent one of the other adverse event outcomes, the important medical event should be reported as serious."

All SAEs that are unexpected and related to the study drug will be reported. The investigator is responsible for informing HSA no later than 15 calendar days after first knowledge that the case qualifies for expedited reporting. Follow-information will be actively sought and submitted as it becomes available. For fatal or life-threatening cases, HSA will be notified as soon as possible but no later than 7 calendar days after first knowledge that a case qualifies, followed by a complete report within 8 additional calendar days.

ELIGIBILITY:
Inclusion Criteria:

1.1. Inclusion Criteria

The obese subject must meet all of the following inclusion criteria to participate in this study:

1. Ideal body weight for height (WFH) of at least 140% or BMI for age above 97th percentile
2. Overweight before 10 years of age
3. Informed consent from both obese children subject and legal representative e.g. parents

Family member must meet all of the following inclusion criteria to participate in this study:

1. Must be parent or direct sibling of obese subject
2. Informed consent from both subject and parent is subject is below 21 years of age

Exclusion Criteria:

All subjects meeting any of the exclusion criteria at baseline will be excluded from participation:

1. Unfit for blood testing and OGTT testing
2. No informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: As our study aims to identify susceptible genetic variants associated with early onset obesity, we will be recruiting 400 obese children to participate in this genetic study, in addition to the existing DNA samples we collected in a previous study. These 400 obese children will be recruited through NUH paediatric clinic and School Health Clinic at Health Promotion Board. We will also recruit family members of the obese children who are interested to join the research study. We will be using the DNA samples and information of 250 obese children previously recruited to the Obesity Genetic Study from January 2000 to December 2004 . We will also be performing WES on 500 lean adults (as controls) recruited for an ongoing study.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Identify novel obesity genes and variants using whole-exome sequencing (WES) in our local Singaporean obese children. | 3 years
  whole exom sequencing data

SECONDARY OUTCOMES:
Assess and compare the metabolic phenotype of the current severely obese children and severely obese children recruited in a similar fashion 15 years ago by the obesity gene study (OGS) group. | 3 years
  metabolic measures
Biomarkers, inflammatory markers and PBMC gene expressions between metabolically healthy obese and metabolically unhealthy obese | 3 years
  Inflammatory measures
Stool microbiota/metagenomics in obese children, and metabolic health | 3 years
  Microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Yung Seng Lee, M.D, PhD, Principal Investigator — National University Health System
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - Health Promotion Board, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng SB, Turner EH, Robertson PD, Flygare SD, Bigham AW, Lee C, Shaffer T, Wong M, Bhattacharjee A, Eichler EE, Bamshad M, Nickerson DA, Shendure J. Targeted capture and massively parallel sequencing of 12 human exomes. Nature. 2009 Sep 10;461(7261):272-6. doi: 10.1038/nature08250. Epub 2009 Aug 16. PMID 19684571
- [Background] Hinney A, Nguyen TT, Scherag A, Friedel S, Bronner G, Muller TD, Grallert H, Illig T, Wichmann HE, Rief W, Schafer H, Hebebrand J. Genome wide association (GWA) study for early onset extreme obesity supports the role of fat mass and obesity associated gene (FTO) variants. PLoS One. 2007 Dec 26;2(12):e1361. doi: 10.1371/journal.pone.0001361. PMID 18159244
- [Background] Ramachandrappa S, Farooqi IS. Genetic approaches to understanding human obesity. J Clin Invest. 2011 Jun;121(6):2080-6. doi: 10.1172/JCI46044. Epub 2011 Jun 1. PMID 21633175